CLINICAL TRIAL: NCT04638439
Title: A Phase Ib, Open Label Study to Assess the Safety and Efficacy of Sequential Administration of P1101 and Anti-PD1 in Interferon-Naive Adults With Chronic Hepatitis B or D Infection
Brief Title: The Safety and Efficacy of Sequential Treatment of Ropeginterferon Alfa-2b (P1101) and Anti-PD1 in Interferon-Naive Adults With Chronic Hepatitis B or D Infection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PharmaEssentia (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A20-101
Record Dates: First submitted 2020-11-06; First posted 2020-11-20 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Chronic Hepatitis B Infection; Chronic Hepatitis D Infection
Keywords: P1101; Anti-PD1; HBV; HDV
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Nivolumab; entecavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- P1101 + Nivolumab + Entecavir (Experimental)
  Interventions: Drug: P1101 + Nivolumab + Entecavir

INTERVENTIONS:
Drug: P1101 + Nivolumab + Entecavir — P1101 (Ropeginterferon alfa-2b) 450 µg subcutaneously (SC) Q2W for 6 doses (12 weeks), followed by 0.3 mg/kg Nivolumab for 6 doses (12 weeks), with a follow up of 24 weeks. All patients will also receive Entecavir 0.5 mg QD from Day 1 to Follow-up 24.
  Other Names: P1101 (Ropeginterferon alfa-2b) + Nivolumab + Entecavir

SUMMARY:
Primary objective:

To evaluate the safety and tolerability of sequential administration of P1101 and anti-PD1 in patient with chronic hepatitis B or D infection

Secondary objectives:

1. To explore HBsAg loss and kinetics during the study period
2. To assess the anti-viral effect during the study period
3. To evaluate the rate of ALT normalization

DETAILED DESCRIPTION:
There are 20 scheduled visits (screening, treatment weeks & follow-up weeks) for patients which include screening visit, TW0 (baseline), TW2, TW4, TW6, TW8, TW10, TW12, TW13, TW15, TW17, TW19, TW21, TW23 (EOT), FW4, FW8, FW12, FW16, FW20 and FW24.

ELIGIBILITY:
Inclusion Criteria:

1. Positive for HBsAg for at least 6 months, either HBeAg (+) or HBeAg (-), and ALT ≤ 10X ULN at screening;
2. Interferon naïve;
3. Quantitative HBsAg Level < 5,000 IU/mL at screening; HBV DNA < 2,000 IU/mL (patients are either under NUC treatment or not);
4. Adults ≥20 years of age; patients who are over 70 years of age must be in generally good health depending upon the Investigator's judgment;
5. Laboratory test results before study entry: WBC ≥ 3,000/mm3; ANC ≥ 1,500/mm3; Platelet ≥ 90,000/mm3; Hemoglobin ≥ 10g/dL; e-GFR ≥ 60mL/min;
6. ECG without clinically significant abnormalities before study entry;
7. Be able to attend all scheduled visits and to comply with all study procedures;
8. Patients with anti-HDV (+) can be enrolled;
9. Patients with fibrosis stage < F3 can be enrolled;
10. Willing to provide written informed consent;

Exclusion Criteria:

1. Clinically significant illness or surgery that might interfere with study participation;
2. Clinically significant vital sign abnormalities or fever [body temperature >38℃]);
3. History of significant alcohol or drug abuse within 6 months prior to the screening visit (alcohol consumption of more than 14 units of alcohol per week [1 Unit = 150 mL of wine, 360 mL of beer, or 45 mL of 40% alcohol]) or refusal to abstain from alcohol or illicit drugs throughout the study;
4. Any history or presence of poorly controlled or clinically significant medical conditions that are not suitable to receive interferon-based treatment, at the discretion of the investigator: major psychiatric (including but not limited to those with severe depression, severe bi-polar disorder, schizophrenia, suicidal ideation or history of suicidal attempt), neurological, cardiovascular (i.e. uncontrolled hypertension, congestive heart failure (≥ NYHA class 2), serious cardiac arrhythmia, significant coronary artery stenosis, unstable angina) or recent stroke or myocardial infarction), pulmonary, hematologic, immunologic, autoimmune diseases, thyroid or other endocrine diseases, metabolic (e.g. diabetes mellitus with HbA1C > 8.0%) or other uncontrolled systemic disease, coagulation disorders or blood dyscrasias;
5. Pregnant patient, female patient or the spouse of male patient, with child-bearing potential who is unwilling or unable to practice adequate contraception, defined as vasectomy in men, tubal ligation in women, or use of condoms and spermicides, or birth control pills, or intrauterine devices throughout the study;
6. History of severe allergic or hypersensitivity reactions, e.g. hypersensitivity to the active substance or to any of the excipients of Ropeginterferon alfa-2b (P1101), bronchospasm, angioedema, asthma, or anaphylaxis;
7. Therapy with any systemic anti-viral treatment, anti-neoplastic, or immunomodulatory treatment (including supraphysiologic doses of steroids and radiation) within 1 month (3 months for those with long elimination half-lives) prior to the first dose of study drug;
8. A depot injection or an implant of any drug within 3 months prior to administration of study medication, other than contraception or hyaluronic acid injections in joints for osteoarthritis;
9. Body organ transplant or taking immunosuppressant;
10. Use investigational drug of other clinical trials within 4 weeks prior to the first dose of the study drug;
11. History of malignancy diagnosed or treated within 5 years prior to screening (except for localized treatment of squamous or non-invasive basal cell skin cancers; cervical carcinoma in situ);
12. History of opportunistic infection (e.g., invasive candidiasis or pneumocystis pneumonia);
13. Serious localized infection (e.g., cellulitis, abscess) or systemic and life-threatening infection (e.g., septicemia) within 3 months prior to screening;
14. Clinically significant medical conditions known to interfere absorption, distribution, metabolism or excretion of the study drugs;
15. Decompensated liver disease, which includes but not limited to the following: total bilirubin≥2 mg/dL (except in Gilbert syndrome), direct bilirubin ≥2X ULN, albumin level < 3.5 g/dL, INR ≥1.5; clinical evidence of ascites, liver decompensation, hepatic encephalopathy, oesophageal varices or cirrhosis as identified by ultrasound or any other examination before study entry;
16. Significant steatohepatitis by ultrasound or other examination at the discretion of investigator;
17. Other form of significant chronic liver diseases, except those mentioned above (e.g. HBV, HDV);
18. Significant or major fundoscopic findings at screening including but not limited to retinal exudates, hemorrhage, detachment, neovascularization, papilledema, optic atrophy, microaneurysms and macular changes;
19. Positive for anti-HIV or anti-HCV;
20. Prior therapy with anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathway;
21. Any contraindication to receiving anti-PD-1 antibody (e.g. active or a history of life-threatening autoimmune conditions, corticosteroids treatment required) or hypersensitivity to the constituents of anti-PD-1 antibody;
22. Patients under monotherapy by telbivudine or any other combination therapy with telbivudine.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-08-17 (Actual); Primary Completion 2025-05-14 (Actual); Study Completion 2025-05-14 (Actual)

PRIMARY OUTCOMES:
Safety: AE/SAE | Through study Follow-up Week 24 (up to 330 days)
  Number of patients with adverse events, including SAEs
Safety: clinically significant abnormalities | Through study Follow-up Week 24 (up to 330 days)
  Number of patients with clinically significant abnormalities, including vital sign, physical examination, electrocardiogram (ECG) and laboratory data

SECONDARY OUTCOMES:
Subjects with HBsAg loss | Treatment Week 12, Treatment Week 23, Follow-up Week 12 and Follow-up Week 24
  The percentage of subjects with HBsAg loss at treatment week 12, 23 and follow up week 12, 24 in the treatment group
Subjects with HBsAg reduction from baseline | Treatment Week 12, Treatment Week 23, Follow-up Week 12 and Follow-up Week 24
  The percentage of subjects with HBsAg reduction from baseline at treatment week 12, 23 and follow up week 12, 24 in the treatment group
Subjects with HBsAg seroconversion | Treatment Week 12, Treatment Week 23, Follow-up Week 12 and Follow-up Week 24
  The percentage of subjects with HBsAg seroconversion at treatment week 12, 23 and follow up week 12, 24 in the treatment group
Subjects with undetectable HBV DNA | Treatment Week 12, Treatment Week 23, Follow-up Week 12 and Follow-up Week 24
  The percentage of subjects with undetectable HBV DNA at treatment week 12, 23 and follow up week 12, 24 in the treatment group
Subjects with ≥ 2 log10 decline from baseline in HDV RNA | Treatment Week 12, Treatment Week 23, Follow-up Week 12 and Follow-up Week 24
  The percentage of subjects with ≥ 2 log10 decline from baseline in HDV RNA at treatment week 12, 23 and follow up week 12, 24 in the treatment group
Subjects with undetectable HDV RNA | Treatment Week 12, Treatment Week 23, Follow-up Week 12 and Follow-up Week 24
  The percentage of subjects with undetectable HDV RNA at treatment week 12, 23 and follow up week 12, 24 in the treatment group
Subjects with ALT normalization | Treatment Week 12, Treatment Week 23, Follow-up Week 12 and Follow-up Week 24
  The percentage of subjects with ALT normalization at treatment week 12, 23 and follow up week 12, 24 in the treatment group

CONTACTS AND LOCATIONS:
Locations (5):
- Taiwan (5):
  - Chia-Yi Christian Hospital, Chiayi City
  - National Taiwan University Hospital, Taipei
  - Taipei Medical University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Memorial Hospital, Linkou, Taoyuan

IPD SHARING:
Plan to Share IPD: No